CLINICAL TRIAL: NCT01965964
Title: Sydney Swallow Questionnaire: Translation of a Questionnaire Relating to the Function of Swallowing and Validation of the German Version
Brief Title: Translation of the Sydney Swallow Questionnaire and Validation of the German Version
Status: Completed | Type: Observational
Sponsor: University of Zurich (Other)
Responsible Party: Sponsor
Other Study IDs: BJ_05_07_2011
Record Dates: First submitted 2013-10-15; First posted 2013-10-18 (Estimated); Last update posted 2015-12-15 (Estimated); Status verified 2015-12

CONDITIONS: Dysphagia
Keywords: Dysphagia, Swallowing functions, Questionnaire in German
MeSH Terms: conditions — Deglutition Disorders | interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Procedure: Questionnaire

SUMMARY:
Translation of a validated questionnaire (SSQ) from english to german and validation of the german version. The SSQ consists of 17 well-structured questions for the assessment and quantification of patient reported difficulties in swallowing function. The tool is specifically designed to evaluate important aspects of swallowing function The questions cover the symptoms related to combinations of variables like the anatomic region, type of dysfunction, and the consistency of swallowed bolus.

ELIGIBILITY:
Inclusion criteria: - patients with diagnosed dysphagia "of any causes"

* sufficient proficiency in german
* voluntary participation

Exclusion criteria: - insufficient knowledge of the german language

* cognitive limitations
* reduced general state of health

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients suffering from Dysphagia for at least half a year
Sampling Method: Non-Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2013-05; Primary Completion 2013-12 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
Percentage of patients able to understand and fill out the german translation of the questionnaire | Baseline
  Establishment of a questionnaire in german to determine patients' swallowing functions.

CONTACTS AND LOCATIONS:
Overall Officials: Joerg E Bohlender, MD, Principal Investigator — University Hospital Zurich, Division of Otorhinolaryngology
Locations (1):
- University Hospital Zurich, Division of Otorhinolaryngology, Zurich, Canton of Zurich, Switzerland